CLINICAL TRIAL: NCT01204892
Title: Postoperative Pain After Laparoscopic Cholecystectomy in Patients Receiving Bilateral Ultrasound-guided Transverse Abdominis Plane Block Compared With Local Anesthetic Infiltration of Trochar Insertion Sites With Ropivacaine 0.5%
Brief Title: Pain After Laparoscopic Cholecystectomy With Bilateral Tranversus Abdominis Plane (TAP) Block Versus Local Anesthetic Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H-27128
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP Block (Active Comparator): Patient will received bilateral ultrasound-guided TAP block with total of 30 ml of ropivacaine 0.5% after induction of general anesthesia
  Interventions: Procedure: TAP Block
- Local infiltration (Active Comparator): 20 ml of Ropivacaine 0.5% will be injected at port sites after induction of general anesthesia. 7 ml each for 10 mm ports, 3 ml each of 5 mm ports
  Interventions: Procedure: Local infiltration

INTERVENTIONS:
Procedure: TAP Block — Patient will received bilateral ultrasound-guided TAP block with total of 30 ml of ropivacaine 0.5% after induction of general anesthesia
  Arms: TAP Block
Procedure: Local infiltration — 20 ml of Ropivacaine 0.5% will be injected at port sites after induction of general anesthesia. 7 ml each for 10 mm ports, 3 ml each of 5 mm ports
  Arms: Local infiltration

SUMMARY:
The purpose if to find out if analgesia with bilateral ultrasound-guided Tranversus Abdominis Plane (TAP) block with Ropivacaine 0.5% is better than analgesia with local infiltration of trochar sites with Ropivacaine 0.5% in patients undergoing laparoscopic cholecystectomy.

Our hypothesis is that in laparoscopic cholecystectomy, bilateral TAP blocks will reduce postoperative pain scores when compared to conventional postoperative pain control with local infiltration of trochar insertion sites.

DETAILED DESCRIPTION:
The purpose if to find out if analgesia with bilateral ultrasound-guided Tranversus Abdominis Plane (TAP) block with Ropivacaine 0.5% is better than analgesia with local infiltration of trochar sites with Ropivacaine 0.5% in patients undergoing laparoscopic cholecystectomy.

Our hypothesis is that in laparoscopic cholecystectomy, bilateral TAP blocks will reduce postoperative pain scores when compared to conventional postoperative pain control with local infiltration of trochar insertion sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages 18-64
2. American Society of Anesthesiology Physical Status I, II or III
3. Inpatients scheduled to undergo laparoscopic cholecystectomy at Ben Taub General Hospital

Exclusion Criteria:

1. Open cholecystectomy - excluded due to increased levels of pain in open procedures
2. Scheduled for ambulatory surgery
3. Renal dysfunction (Serum Cr > 1.2) - excluded due to potential altered metabolism of anesthetic and pain medications
4. Coagulopathy or anticoagulation - increased risk of bleeding from nerve block injection
5. Allergy or contraindication to any of the study medications or anesthetic agents
6. Chronic opioid analgesic use at home - excluded due to potential difficulty in assessing pain caused by the procedure alone
7. Patient inability to properly describe postoperative pain to investigators (language barrier, dementia, delirium, psychiatric disorder)
8. Pregnancy
9. Prisoners
10. Patient or surgeon refusal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours
  Pain scores on NAS scale (0-10) at the following times:
  Preop, Time 0, Time 1, Time 2, Time 4, Time 8, Time 12, Time 24

SECONDARY OUTCOMES:
PONV (Postoperative nausea and vomiting) | 24 hours
  PONV events in first 24 hours
Narcotics use | 24 hours
  Fentanyl, morphine, and hydrocodone/apap total for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ortiz, MD, Principal Investigator — Batylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States